CLINICAL TRIAL: NCT05920044
Title: The Effects of an Individualized Balance and Proprioception Training Program on Pain and Function in Patients With Chronic Ankle Sprains: A Randomized Controlled Trial
Brief Title: Balance and Proprioception Training Program in Patients With Chronic Ankle Sprains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/Ank-01200021
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: (Experimental): Participants will receive an eight-week individualized balance and proprioception training program.
  Interventions: Other: balance and proprioception training program.
- Control group (Active Comparator): Participants will continue their usual care, including general strength and flexibility exercises.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: balance and proprioception training program. — The program will include exercises focused on improving ankle stability and joint position sense, such as single-leg stance, wobble board, and resistance band exercises.
  Participants will attend two supervised sessions per week and perform home-based exercises 3-4 times per week.
  Progression of exercises will be individualized based on participant performance and tolerance.
  Arms: Intervention Group:
Other: Usual care — Participants will continue their usual care, including general strength and flexibility exercises.
  No specific balance and proprioception training will be provided.
  Arms: Control group

SUMMARY:
To examine the effects of an individualized balance and proprioception training program on pain, function, and the risk of recurrent ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 years
* History of at least two ankle sprains within the last 12 months
* Presence of ankle instability symptoms, such as recurrent giving way or chronic pain

Exclusion Criteria:

* Acute ankle injury within the last six weeks
* Lower extremity fracture within the last six months
* Other musculoskeletal or neurological disorders affecting the lower extremity
* Inability to comply with study requirements

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-27 (Estimated); Primary Completion 2024-06-27 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity | Changes in Pain intensity at baseline, 8 weeks, and 16 weeks follow up
  Pain intensity will be measured using the Numeric Pain Rating Scale (NPRS)
Changes in Functional Ability | Changes in Functional ability at baseline, 8 weeks, and 16 weeks follow up
  Functional ability will be assessed using the Foot and Ankle Ability Measure (FAAM)

SECONDARY OUTCOMES:
Changes in Balance | Changes in balance at baseline, 8 weeks, and 16 weeks follow up
  Balance will be assessed using the Star Excursion Balance Test (SEBT)
Changes in Proprioception | Changes in proprioception at baseline, 8 weeks, and 16 weeks follow up
  Proprioception will be measured using the joint position sense test with an ankle electrogoniometer
Incidence of Recurrent Ankle Sprains | From post-intervention at 8 weeks to the end of the follow-up period at 16 weeks
  Incidence of recurrent ankle sprains during the follow-up period will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No